CLINICAL TRIAL: NCT01139918
Title: Exploratory Study on Quality of Life in Patient With Moderate Psoriasis and Moderate Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: Inno-6017
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Psoriatic Arthritis; Psoriasis
Keywords: psoriatic arthritis; psoriasis; Quality of life
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort A: 40 patients with moderate psoriatic arthritis and moderate psoriasis
- Cohort B: 40 patients with mild psoriatic arthritis and moderate psoriasis
- Cohort C: 40 patients with moderate psoriatic arthritis and mild psoriasis

SUMMARY:
This exploratory study will be used to identify questions that will be part of a new QoL questionnaire for patients with psoriasis and psoriatic arthritis and to determine the sample size needed for its validation. The new questionnaire will be a global QoL questionnaire which will take into account the impact of both psoriasis and psoriatic arthritis on QoL.

STUDY OBJECTIVES

* To evaluate the influence of psoriasis and psoriatic arthritis on patient's answers to QoL questions from DLQI, HAQ, EQ-5D, FACIT-fatigue and SF-36.
* To identify an equal number of questions from DLQI, HAQ, EQ-5D, FACIT-fatigue and SF-36 where answers are mostly influenced either by psoriatic arthritis or by psoriasis.

DETAILED DESCRIPTION:
This study will recruit three cohorts of 40 patients each: moderate psoriatic arthritis and moderate psoriasis, mild psoriatic arthritis and moderate psoriasis, moderate psoriatic arthritis and mild psoriasis. Eligible patients will fill the following questionnaires: Dermatology Life Quality Index (DLQI), Health Assessment Questionnaire (HAQ), EQ-5D, Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-fatigue) and 36-Item Short Form Health Survey Questionnaire (SF-36). In addition, each patient will be asked on a 4 point Likert scale how much their answer to each question is related to the impact of their skin disease or their psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with plaque psoriasis and psoriatic arthritis with either:

  * Moderate psoriatic arthritis and moderate psoriasis defined as: [psoriatic arthritis with either 3-7 joints showing signs of synovitis OR a BASDAI of 2-4] AND [between 3 to less than 10% of the body surface area involved with psoriasis] (COHORT A) OR
  * Mild psoriatic arthritis and Moderate psoriasis defined as: [psoriatic arthritis with either 1-2 joints showing signs of synovitis OR a BASDAI greater than 0 but less than 2] AND [between 3 to less than 10% of the body surface area involved with psoriasis] (COHORT B) OR
  * Moderate psoriatic arthritis and Mild psoriasis defined as: [psoriatic arthritis with either 3-7 joints showing signs of synovitis OR a BASDAI of 2-4] AND [more than 0 but less than 3% of the body surface area involved with psoriasis] (COHORT C)
* Patient is between 18 years and older.
* Patient is capable of reading and understanding French or English questionnaires.
* Patient is capable of giving informed consent.

Exclusion Criteria:

* Patient has presence of eythrodermic, pustular or guttate psoriasis.
* Patient has another non psoriatic arthropathy (such as osteoarthritis) that could have a significant impact of QoL related to psoriatic arthritis
* Patient has another non psoriatic dermatosis that could have a significant impact on QoL related to psoriasis
* Patient has any other co-morbidity with a severity that could have a significant impact on QoL
* Patient has had a significant flare-up of psoriasis or psoriatic arthritis within 90 days of Day 0
* Patient has received investigational drugs within four weeks prior to Day 0
* Patient has been treated with systemic anti-psoriatic drugs such as steroids, retinoids, cyclosporine, PUVA therapy within the four weeks prior to Day 0. Methotrexate, sulphasalazine and leflunomide are allowed during the study as long as patient has been on a stable dose within 90 days of Day 0.
* Patient has been treated with ultraviolet light therapy (UVB, nbUVB) within the two weeks prior to Day 0
* Patient has used biologics (such etanercept, adalimumab, infliximab, abatacept, ustekinumab) within 180 days of Day 0
* Patient is currently pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study popululation description: Patients suffering from either: moderate psoriatic arthritis and moderate psoriasis, mild psoriatic arthritis and moderate psoriasis or moderate psoriatic arthritis and mild psoriasis, known from dermatologists participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2010-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
There is no primary outcome in this study. See objectives. | 1 Day
  There is no primary outcome in this study. Patients with psoriatic arthritis and psoriasis answer questionnaires on one occasion.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (10):
- Canada (10):
  - Kirk Barber Research, Calgary, Alberta
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Dermatrials Research, Hamilton, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Quebec
  - Clinique Médicale Dr Isabelle Delorme, Saint-Hyacinthe, Quebec
  - Diex Research Sherbrooke east, Sherbrooke, Quebec